CLINICAL TRIAL: NCT00365027
Title: Transfer of Fresh Versus Frozen/Thawed Embryos in IVF Cycles Where GnRH Agonist is Utilized for Oocyte Maturation.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5040706
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Ovarian Hyperstimulation Syndrome; Infertility Drugs; Female
Keywords: GNRH agonist; ovarian hyperstimulation syndrome; Embryo cryopreservation
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

INTERVENTIONS:
Procedure: Delayed embryo transfer

SUMMARY:
It has been suggested that in IVF cycles where GNRH agonist is utilized for final oocyte maturation in patients at risk of ovarian hyperstimulation, pregnancy rates are reduced. We hypothesize that the use of GNRH antagonist reduces pregnancy rates through an effect on the endometrium and not oocyte quality, therefore better results may be obtained by not returning these embryos in a fresh cycle but rather cryopreserving them and returning them to the uterus and a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Woman at risk of ovarian hyperstimulation syndrome in IVF cycles for whom GNRH agonist was utilized for final oocyte maturation

Exclusion Criteria:

* Patient's refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Implantation rate per transfer
Pregnancy rate per embryo transfer
Implantation rate per IVF cycle
Pregnancy rate per IVF cycle

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Shalev, Study Chair — HaE'mek medical center